CLINICAL TRIAL: NCT03957915
Title: A Phase I, First in Human, Open-label Study of Escalating Doses of INA03 Administered Intravenously as Single Agent in Adult Patients With Relapse/Refractory Acute Leukemia
Brief Title: Study of Escalating Doses of INA03 Administered Intravenously as Single Agent in Adult Patients With Relapse/Refractory Acute Leukemia
Acronym: INA03
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: INATHERYS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INA03-IPC 2018-008; 2019-000814-13 (EudraCT Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia Recurrent; Acute Lymphoblastic Leukemia, in Relapse; Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukaemia Recurrent; Mixed Phenotype Acute Leukemia
Keywords: acute leukemia; refractory; in relapse; antibody drug conjugate; first in human; escalating doses; INA03
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute

STUDY DESIGN:
Intervention Model Description: This Phase 1 Study is an open-label, non-randomized, dose escalation, safety, efficacy, pharmacokinetic, and pharmacodynamic evaluation study of INA03 administered as a single agent IV infusion every 2 weeks to patients ≥18 years of age with R/R AML, MLL, or ALL.
  The study will be performed in 2 parts: a Dose Titration for Day 1 study (Part 1) followed by a Dose Escalation Part (Part 2) of INA03 used as monotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INA03 (Experimental): INA03 administration
  Interventions: Drug: INA03 administration

INTERVENTIONS:
Drug: INA03 administration — INA03 will be administered IV on Day 1, Day 14 of 28-day cycles. The administration of INA03 will begin at 0.02 mg/kg. Study Part I is a titration study to determine the dose for the first INA03 infusion. Patients will be enrolled in sequential cohorts of 2 patients to receive ascending starting doses of INA03, starting from the lowest starting dose (0.02 mg/kg), and followed by subsequent administrations of INA03 (D14 and beyond) at a fixed dose of 0.1 mg/kg. The starting dose will be increased every cohort of 2 patients until evidence of absence of marrow residual erythroblasts by D14 myelogram. This dose is referred to as the MEID and will be selected as the D1 dose for the study Part 2. Patient accumulation in Part I of the study will continue until no evidence of non-hematological DLT within 28 days post dosing

SUMMARY:
This Phase 1 Study is an open-label, non-randomized, dose escalation, safety, efficacy, pharmacokinetic, and pharmacodynamic evaluation study of INA03 administered as a single agent IV infusion every 2 weeks to patients ≥18 years of age with R/R AML, MLL, or ALL.

The study will be performed in 2 parts: a Dose Titration for Day 1 study (Part 1) followed by a Dose Escalation Part (Part 2) of INA03 used as monotherapy.

DETAILED DESCRIPTION:
This Phase 1 Study is an open-label, non-randomized, dose escalation, safety, efficacy, pharmacokinetic, and pharmacodynamic evaluation study of INA03 administered as a single agent IV infusion every 2 weeks to patients ≥18 years of age with R/R AML, MLL, or ALL.

The study will be performed in 2 parts: a Dose Titration for Day 1 study (Part 1) followed by a Dose Escalation Part (Part 2) of INA03 used as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

. Patient with

* cytologically confirmed and documented B-cell or T-cell ALL or de novo, secondary or therapy-related AML or Mixed Phenotype Acute Leukemia (MPAL) defined according to World Health Organization (WHO) 2016 classification28 AND
* with 20% or more CD71 positive blast cells
* in relapse after- or refractory to registered therapies or ineligible to standard treatments
* with circulating blasts ≤ 20 000/mm3. For eligible patients with AML/ALL with blasts > 20000/mm3, a treatment with hydroxyurea is allowed to maintain tumor cells ≤ 20000/mm3 2. Male or female age ≥ 18 years 3. WHO performance status 0-2 4. Following laboratory values unless considered due to the leukemia:

  1. AST and or ALT ≤ 2.5 ULN
  2. Total bilirubin level < 1.5 ULN (except Gilbert disease)
  3. Serum creatinine ≤ 1.5 ULN
  4. LDH < 3-5 ULN
  5. Uric acid ≤8 mg/dl
  6. Electrolyte panel within normal range
  7. Urine Dipstick Reading negative for proteinuria or, if documentation of +1 results for protein on dipstick reading, then total urinary protein ≤ 500 mg and measured creatinine clearance ≥50mL/min/1.73m2 from a 24-hour urine collection
  8. Patients who have recovered at least CTCAE grade <2 5. Life expectancy greater than 3 months 6. Women of child bearing potential must be willing to use birth control method during the study duration (W4 or early termination) plus 30 days. Male partner of women must use condom; in case of male patient, he must agree to use condom during the study duration (W4 or early termination) plus 30 days; 7. Pregnancy test (females of childbearing potential): negative 8. Signed informed consent indicating that they have been informed of the procedures to be followed, an is willing and able to comply the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts 9. Patient affiliated to the national "Social Security" regimen or beneficiary of this regi-men

     Exclusion Criteria:
     1. Patients with acute promyelocytic leukemia
     2. Patients with more than 30% marrow erythroid cells
     3. Patients who have been treated with any anti-TfR antibody
     4. Allogeneic stem cell transplantation in the last 6 months or with persistent active GVHD. Autologous bone marrow transplant in the last 3 months
     5. Last dose of prior chemotherapy, immunotherapy or investigational agent within 14 days or within 5 half-lives before baseline receipt of study medication, except for hydroxyurea and corticosteroids

     7. Patients who have had a prior anaphylactic or other severe infusion reaction such that the patient is unable to tolerate human immunoglobulin or monoclonal antibody administration 8. Patients who have history or clinical evidence of central nervous system (CNS), meningeal, or epidural disease from any cause and/or peripheral neuropathy 9. Impaired cardiac function or clinically significant cardiac disease, including any one of the following:

  a. New York Heart Association Class III or IV cardiac disease, including preexisting clinically significant arrhythmia, congestive heart failure, or cardiomyopathy b. Angina pectoris ≤ 3 months prior to starting study drug c. Acute myocardial infarction ≤ 3 months prior to starting study drug d. Other clinically significant heart disease (e.g., uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen) e. Left ventricular Ejection Fraction <45% 11. Uncontrolled infection 12. Acute and chronic liver disease 13. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnor-mality that may increase the risk associated with study participation or study drug administra-tion or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study.

  14. Patients with prior radiation therapy
  1. ≤12 weeks for cranial radiation therapy
  2. ≤ 4 weeks for wide field radiation therapy
  3. ≤2 weeks for involved field radiation therapy 15. Major surgery ≤ 4weeks prior to starting study drug or who have not recovered from side effects of such therapy 16. Known diagnosis of HIV infection (HIV testing is not mandatory). 17. History of another primary malignancy that is currently clinically significant or currently requires active intervention 18. Pregnant or breastfeeding patient; 19. Active drug or alcohol dependence; 20. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Determination of the minimal erythroblastopenia-inducing dose (MEID) for INA03 in adults with refractory/relapsed acute leukemia | within 2 weeks from initial dosing
  MEID defined as the lowest dose associated with the risks of residual erythroblasts in the bone marrow at 2 weeks from initial dosing or grade 2 or above non hematologic toxicity within 2 weeks from initial dosing
Determination of the maximum tolerated dose (MTD) for subsequent administrations (D15 from initial dosing and beyond) for INA03 in adults with refractory/relapsed acute leukemia | 28 days from the first administration of INA03
  the maximum tolerated dose (MTD) for subsequent administrations (D15 from initial dosing and beyond)

SECONDARY OUTCOMES:
Safety of INA03: NCI-CTCAE v5.0 | Until 30 days after last dose
  Safety from the findings of reports of adverse events based on incidence, severity (as graded by the NCI-CTCAE v5.0), cumulative nature of treatment-emergent adverse event (TEAEs)
pharmacokinetic (PK) profile of INA03 | From initial dosing day to Day 42
  Peak Plasma Concentration (Cmax) will be calculated, as appropriate
pharmacokinetic (PK) profile of INA03 | From initial dosing day to Day 42
  Area under the plasma concentration versus time curve (AUC) will be calculated, as appropriate
pharmacokinetic (PK) profile of INA03 | From initial dosing day to Day 42
  The terminal half-life will be calculated, as appropriate
pharmacodynamics (PD) profile of INA03 | From screening to end of study visit (maximum 182 days)
  PD according to variation of erythroblast and blasts decrease using bone marrow as-pirate (BMA), and blood samples before and under treatment
Concentration of anti-INA03 antibodies | From screening to end of study visit (maximum 182 days)
  Serum concentration of anti-INA03 antibodies in micrograms per milliliter
Preliminary clinical response of INA03 | from the date of treatment initiation (Day-1) to the date of relapse, progression or death, whichever comes first (a maximum 182 days)
  Clinical response as defined by European LeukemiaNet (ELN) 2017 recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Norbert VEY, Pr, Principal Investigator — Institut Paoli-Calmettes
Locations (3):
- France (3):
  - Institut Paoli-Calmettes, Marseille, Bouches-du Rhône
  - Chu Bordeaux Hopital Haut Leveque, Pessac
  - IUCT, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kell J. Considerations and challenges for patients with refractory and relapsed acute myeloid leukaemia. Leuk Res. 2016 Aug;47:149-60. doi: 10.1016/j.leukres.2016.05.025. Epub 2016 Jun 11. PMID 27371910
- [Background] Dohner H, Dolnik A, Tang L, Seymour JF, Minden MD, Stone RM, Del Castillo TB, Al-Ali HK, Santini V, Vyas P, Beach CL, MacBeth KJ, Skikne BS, Songer S, Tu N, Bullinger L, Dombret H. Cytogenetics and gene mutations influence survival in older patients with acute myeloid leukemia treated with azacitidine or conventional care. Leukemia. 2018 Dec;32(12):2546-2557. doi: 10.1038/s41375-018-0257-z. Epub 2018 Oct 1. PMID 30275526
- [Background] Eleni LD, Nicholas ZC, Alexandros S. Challenges in treating older patients with acute myeloid leukemia. J Oncol. 2010;2010:943823. doi: 10.1155/2010/943823. Epub 2010 Jun 10. PMID 20628485
- [Background] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659
- [Background] Breems DA, Lowenberg B. Acute myeloid leukemia and the position of autologous stem cell transplantation. Semin Hematol. 2007 Oct;44(4):259-66. doi: 10.1053/j.seminhematol.2007.08.002. PMID 17961725
- [Background] Stone RM, Mandrekar SJ, Sanford BL, Laumann K, Geyer S, Bloomfield CD, Thiede C, Prior TW, Dohner K, Marcucci G, Lo-Coco F, Klisovic RB, Wei A, Sierra J, Sanz MA, Brandwein JM, de Witte T, Niederwieser D, Appelbaum FR, Medeiros BC, Tallman MS, Krauter J, Schlenk RF, Ganser A, Serve H, Ehninger G, Amadori S, Larson RA, Dohner H. Midostaurin plus Chemotherapy for Acute Myeloid Leukemia with a FLT3 Mutation. N Engl J Med. 2017 Aug 3;377(5):454-464. doi: 10.1056/NEJMoa1614359. Epub 2017 Jun 23. PMID 28644114
- [Background] Perl AE, Altman JK, Cortes J, Smith C, Litzow M, Baer MR, Claxton D, Erba HP, Gill S, Goldberg S, Jurcic JG, Larson RA, Liu C, Ritchie E, Schiller G, Spira AI, Strickland SA, Tibes R, Ustun C, Wang ES, Stuart R, Rollig C, Neubauer A, Martinelli G, Bahceci E, Levis M. Selective inhibition of FLT3 by gilteritinib in relapsed or refractory acute myeloid leukaemia: a multicentre, first-in-human, open-label, phase 1-2 study. Lancet Oncol. 2017 Aug;18(8):1061-1075. doi: 10.1016/S1470-2045(17)30416-3. Epub 2017 Jun 20. PMID 28645776
- [Background] DiNardo CD, Stein EM, de Botton S, Roboz GJ, Altman JK, Mims AS, Swords R, Collins RH, Mannis GN, Pollyea DA, Donnellan W, Fathi AT, Pigneux A, Erba HP, Prince GT, Stein AS, Uy GL, Foran JM, Traer E, Stuart RK, Arellano ML, Slack JL, Sekeres MA, Willekens C, Choe S, Wang H, Zhang V, Yen KE, Kapsalis SM, Yang H, Dai D, Fan B, Goldwasser M, Liu H, Agresta S, Wu B, Attar EC, Tallman MS, Stone RM, Kantarjian HM. Durable Remissions with Ivosidenib in IDH1-Mutated Relapsed or Refractory AML. N Engl J Med. 2018 Jun 21;378(25):2386-2398. doi: 10.1056/NEJMoa1716984. Epub 2018 Jun 2. PMID 29860938
- [Background] Castaigne S, Pautas C, Terre C, Raffoux E, Bordessoule D, Bastie JN, Legrand O, Thomas X, Turlure P, Reman O, de Revel T, Gastaud L, de Gunzburg N, Contentin N, Henry E, Marolleau JP, Aljijakli A, Rousselot P, Fenaux P, Preudhomme C, Chevret S, Dombret H; Acute Leukemia French Association. Effect of gemtuzumab ozogamicin on survival of adult patients with de-novo acute myeloid leukaemia (ALFA-0701): a randomised, open-label, phase 3 study. Lancet. 2012 Apr 21;379(9825):1508-16. doi: 10.1016/S0140-6736(12)60485-1. Epub 2012 Apr 5. PMID 22482940
- [Background] Cortes JE, Heidel FH, Hellmann A, Fiedler W, Smith BD, Robak T, Montesinos P, Pollyea DA, DesJardins P, Ottmann O, Ma WW, Shaik MN, Laird AD, Zeremski M, O'Connell A, Chan G, Heuser M. Randomized comparison of low dose cytarabine with or without glasdegib in patients with newly diagnosed acute myeloid leukemia or high-risk myelodysplastic syndrome. Leukemia. 2019 Feb;33(2):379-389. doi: 10.1038/s41375-018-0312-9. Epub 2018 Dec 16. PMID 30555165
- [Background] Vey N, Keating M, Giles F, Cortes J, Beran M, Estey E. Effect of complete remission on survival in patients with acute myelogenous leukemia receiving first salvage therapy. Blood. 1999 May 1;93(9):3149-50. No abstract available. PMID 10336269
- [Background] Estey EH. Treatment of relapsed and refractory acute myelogenous leukemia. Leukemia. 2000 Mar;14(3):476-9. doi: 10.1038/sj.leu.2401568. PMID 10720145
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Rowe JM, Buck G, Burnett AK, Chopra R, Wiernik PH, Richards SM, Lazarus HM, Franklin IM, Litzow MR, Ciobanu N, Prentice HG, Durrant J, Tallman MS, Goldstone AH; ECOG; MRC/NCRI Adult Leukemia Working Party. Induction therapy for adults with acute lymphoblastic leukemia: results of more than 1500 patients from the international ALL trial: MRC UKALL XII/ECOG E2993. Blood. 2005 Dec 1;106(12):3760-7. doi: 10.1182/blood-2005-04-1623. Epub 2005 Aug 16. PMID 16105981
- [Background] O'Brien S, Schiller G, Lister J, Damon L, Goldberg S, Aulitzky W, Ben-Yehuda D, Stock W, Coutre S, Douer D, Heffner LT, Larson M, Seiter K, Smith S, Assouline S, Kuriakose P, Maness L, Nagler A, Rowe J, Schaich M, Shpilberg O, Yee K, Schmieder G, Silverman JA, Thomas D, Deitcher SR, Kantarjian H. High-dose vincristine sulfate liposome injection for advanced, relapsed, and refractory adult Philadelphia chromosome-negative acute lymphoblastic leukemia. J Clin Oncol. 2013 Feb 20;31(6):676-83. doi: 10.1200/JCO.2012.46.2309. Epub 2012 Nov 19. PMID 23169518
- [Background] Faderl S, Thomas DA, O'Brien S, Ravandi F, Garcia-Manero G, Borthakur G, Ferrajoli A, Verstovsek S, Ayoubi M, Rytting M, Feliu J, Kantarjian HM. Augmented hyper-CVAD based on dose-intensified vincristine, dexamethasone, and asparaginase in adult acute lymphoblastic leukemia salvage therapy. Clin Lymphoma Myeloma Leuk. 2011 Feb;11(1):54-9. doi: 10.3816/CLML.2011.n.007. PMID 21454191
- [Background] Kolb HJ, Simoes B, Schmid C. Stem cell transplants for patients with relapsed/refractory leukaemia. Curr Opin Hematol. 2009 Nov;16(6):444-52. doi: 10.1097/MOH.0b013e3283309647. PMID 19652599
- [Background] Wolach O, Stone RM. How I treat mixed-phenotype acute leukemia. Blood. 2015 Apr 16;125(16):2477-85. doi: 10.1182/blood-2014-10-551465. Epub 2015 Jan 20. PMID 25605373
- [Background] Lepelletier Y, Camara-Clayette V, Jin H, Hermant A, Coulon S, Dussiot M, Arcos-Fajardo M, Baude C, Canionni D, Delarue R, Brousse N, Benaroch P, Benhamou M, Ribrag V, Monteiro RC, Moura IC, Hermine O. Prevention of mantle lymphoma tumor establishment by routing transferrin receptor toward lysosomal compartments. Cancer Res. 2007 Feb 1;67(3):1145-54. doi: 10.1158/0008-5472.CAN-06-1962. PMID 17283149
- [Background] Daniels-Wells TR, Penichet ML. Transferrin receptor 1: a target for antibody-mediated cancer therapy. Immunotherapy. 2016 Sep;8(9):991-4. doi: 10.2217/imt-2016-0050. Epub 2016 Jul 4. No abstract available. PMID 27373880
- [Background] Ryschich E, Huszty G, Knaebel HP, Hartel M, Buchler MW, Schmidt J. Transferrin receptor is a marker of malignant phenotype in human pancreatic cancer and in neuroendocrine carcinoma of the pancreas. Eur J Cancer. 2004 Jun;40(9):1418-22. doi: 10.1016/j.ejca.2004.01.036. PMID 15177502
- [Background] Callens C, Moura IC, Lepelletier Y, Coulon S, Renand A, Dussiot M, Ghez D, Benhamou M, Monteiro RC, Bazarbachi A, Hermine O. Recent advances in adult T-cell leukemia therapy: focus on a new anti-transferrin receptor monoclonal antibody. Leukemia. 2008 Jan;22(1):42-8. doi: 10.1038/sj.leu.2404958. Epub 2007 Sep 27. PMID 17898788
- [Background] Kolodych S, Koniev O, Baatarkhuu Z, Bonnefoy JY, Debaene F, Cianferani S, Van Dorsselaer A, Wagner A. CBTF: new amine-to-thiol coupling reagent for preparation of antibody conjugates with increased plasma stability. Bioconjug Chem. 2015 Feb 18;26(2):197-200. doi: 10.1021/bc500610g. Epub 2015 Jan 23. PMID 25614935
- [Background] Saber H, Gudi R, Manning M, Wearne E, Leighton JK. An FDA oncology analysis of immune activating products and first-in-human dose selection. Regul Toxicol Pharmacol. 2016 Nov;81:448-456. doi: 10.1016/j.yrtph.2016.10.002. Epub 2016 Oct 13. PMID 27743776
- [Background] Malleret B, Xu F, Mohandas N, Suwanarusk R, Chu C, Leite JA, Low K, Turner C, Sriprawat K, Zhang R, Bertrand O, Colin Y, Costa FT, Ong CN, Ng ML, Lim CT, Nosten F, Renia L, Russell B. Significant biochemical, biophysical and metabolic diversity in circulating human cord blood reticulocytes. PLoS One. 2013 Oct 8;8(10):e76062. doi: 10.1371/journal.pone.0076062. eCollection 2013. PMID 24116088
- [Background] Liu Q, Wang M, Hu Y, Xing H, Chen X, Zhang Y, Zhu P. Significance of CD71 expression by flow cytometry in diagnosis of acute leukemia. Leuk Lymphoma. 2014 Apr;55(4):892-8. doi: 10.3109/10428194.2013.819100. Epub 2013 Aug 20. PMID 23962073
- [Background] Wu B, Shi N, Sun L, Liu L. Clinical value of high expression level of CD71 in acute myeloid leukemia. Neoplasma. 2016;63(5):809-15. doi: 10.4149/neo_2016_519. PMID 27468886
- [Background] Mathis S, Chapuis N, Debord C, Rouquette A, Radford-Weiss I, Park S, Dreyfus F, Lacombe C, Bene MC, Kosmider O, Fontenay M, Bardet V. Flow cytometric detection of dyserythropoiesis: a sensitive and powerful diagnostic tool for myelodysplastic syndromes. Leukemia. 2013 Oct;27(10):1981-7. doi: 10.1038/leu.2013.178. Epub 2013 Jun 14. PMID 23765225
- [Background] Suzuki N, Suwabe N, Ohneda O, Obara N, Imagawa S, Pan X, Motohashi H, Yamamoto M. Identification and characterization of 2 types of erythroid progenitors that express GATA-1 at distinct levels. Blood. 2003 Nov 15;102(10):3575-83. doi: 10.1182/blood-2003-04-1154. Epub 2003 Jul 31. PMID 12893747
- [Background] Younes A, Bartlett NL, Leonard JP, Kennedy DA, Lynch CM, Sievers EL, Forero-Torres A. Brentuximab vedotin (SGN-35) for relapsed CD30-positive lymphomas. N Engl J Med. 2010 Nov 4;363(19):1812-21. doi: 10.1056/NEJMoa1002965. PMID 21047225
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Han TH, Gopal AK, Ramchandren R, Goy A, Chen R, Matous JV, Cooper M, Grove LE, Alley SC, Lynch CM, O'Connor OA. CYP3A-mediated drug-drug interaction potential and excretion of brentuximab vedotin, an antibody-drug conjugate, in patients with CD30-positive hematologic malignancies. J Clin Pharmacol. 2013 Aug;53(8):866-77. doi: 10.1002/jcph.116. Epub 2013 Jun 10. PMID 23754575